CLINICAL TRIAL: NCT01390181
Title: The Effect of Losartan Treatment on Matrix Metalloproteinase Levels and Outcomes in Bicuspid Aortic Valve Patients
Brief Title: The Effect of Losartan in Bicuspid Aortic Valve Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment the decision was made to terminate study prior to final data collection for any individual.
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Anna Booher, MD, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00048364
Record Dates: First submitted 2011-06-30; First posted 2011-07-08 (Estimated); Results first posted 2017-04-14 (Actual); Last update posted 2017-04-14 (Actual); Status verified 2017-03

CONDITIONS: Bicuspid Aortic Valve; Thoracic Aortic Aneurysm
MeSH Terms: conditions — Bicuspid Aortic Valve Disease; Aortic Aneurysm, Thoracic | interventions — Losartan

ARMS (1):
- Losartan (Experimental)
  Interventions: Drug: Cozaar

INTERVENTIONS:
Drug: Cozaar — Angiotensin II Receptor Blocker
  Other Names: Losartan

SUMMARY:
The specific aims of this study are to:

* Establish baseline levels of circulating MMP-2 and -9 , TIMP-1and- 2 and TGFB levels in individuals with bicuspid aortic valve and ascending aortic or aortic sinus measurements >40mm.
* Assess the effect on MMP levels during treatment with losartan, an angiotensin II receptor blocking agent.
* In the setting of losartan therapy for one year, evaluate the response of MMP levels in these patients, and clinical outcomes including effects on aortic growth rate

ELIGIBILITY:
Inclusion Criteria:

* Adults >age 18 years and < 65 years old
* Able to give informed consent
* Presence of a bicuspid aortic valve (functional or true bicommisural)and ascending aorta or sinus of Valsalva >4.0cm
* No contraindications to treatment with Losartan, an Angiotensin II receptor blocker
* Able to safely participate in a 4 week drug washout period if currently taking an angiotensin II receptor blocker or ACE inhibitor.

Exclusion Criteria:

* Unable to safely take losartan due to one or more of the following:

  * Hypersensitivity to losartan or other angiotensin receptor blockers
  * Pregnancy
  * Nursing mothers
  * History of angioedema
  * Hypotension - chronically volume depleted patients
  * Hepatic or renal impairment (Cr>1.5mg/dL)
  * Hyperkalemia (K+>4.8)
  * Renal artery stenosis
  * Severe congestive heart failure (class III-IV)
  * Currently taking potassium supplements or salt substitutes containing potassium
  * Currently taking lithium
* Prior surgical intervention to aorta or aortic valve
* Unable or unwilling to give informed consent and follow up with study activities
* Currently taking an angiotensin receptor blocker or ACE inhibitor specifically for hypertension and are therefore unable to or are unwilling to participate in a 4 week drug washout period.
* Females of child bearing who are unwilling to practice adequate birth control throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2011-09; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Booher, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan
Started | 4
Completed | 0
Not Completed | 4
Not completed — Lost to Follow-up | 1
Not completed — Study Terminated due to Low Accrual | 3

BASELINE CHARACTERISTICS:
Arm/Group | Losartan
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Inflammatory Markers Levels
Description: Changes in levels of Matrix Metalloproteinase (MMP-2, MMP-9), Tissue Inhibitor of Metalloproteinases (TIMP 1, TIMP 2), & Transforming Growth Factor-Beta (TGFB) in circulation while taking medication from baseline at 3 months, 6 months and 12 months. The 12 month levels were the primary outcome.
Time Frame: Baseline and 12 months
Population: No participants were analyzed because the study terminated prior to data collection for final primary outcome measure.
Arm/Group | Losartan
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 6 months (study was terminated prior to proposed completion)
Arm/Group | Losartan
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 2/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=4)
Increase in Blood Pressure (Cardiac disorders) | 1 (1)
Shingles (Nervous system disorders) | 1 (1)
Cardiace Disorder (Cardiac disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fall (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes